CLINICAL TRIAL: NCT00376246
Title: Effect of Ezetimibe on Flow-mediated Brachial Artery Reactivity in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ori Ben-Yehuda, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 050714
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Endothelial Dysfunction
MeSH Terms: interventions — Ezetimibe

ARMS (2):
- Group 1 (Other): 1st group will receive Ezetimibe for 2 weeks followed by washout (no medication) period for 4 weeks and followed by placebo for 2 weeks.
  Interventions: Drug: Ezetimibe
- Group 2 (Other): 2nd group will receive Ezetimibe and placebo in reverse order with interspaced 4-week washout period.
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe

SUMMARY:
The objective of this study is to show that Ezetimibe will improve endothelial function following high cholesterol meals in healthy subjects by decreasing absorption of cholesterol and thus affecting concentration and composition of remnant-like particles.

DETAILED DESCRIPTION:
24 subjects will be recruited. Exclusion criteria will be presence of known metabolic syndrome as well as history of coronary artery disease, hypertension, diabetes, cardiomyopathy and tobacco use. Study will be conducted as double blind placebo controlled crossover trial. Subjects will be randomized to 2 groups. 1st group will receive Ezetimibe for 2 weeks followed by washout (no medication) period for 4 weeks and followed by placebo for 2 weeks. 2nd group will receive Ezetimibe and placebo in reverse order with interspaced 4-week washout period. Each subject will be evaluated during 2 visits at the ends of the intervention periods (Ezetimibe and placebo). Visits will occur after 2 and 8 weeks after enrollment. Subjects will be asked to fast 12 hrs before each visit. During each visit, a subject will undergo brachial artery reactivity study (BART) before consumption of standardized high cholesterol meal and at 3 and 6-hour points after the meal. The standardized high cholesterol meal will consist of 2 Egg McMuffin® sandwiches. This meal weighs 276 g and contains 34g of protein, 60g of carbohydrates, 22g of total fat and 470 mg of cholesterol and has 290 Calories. Subjects also will have blood draws for serum lipid measurement performed before each BART procedure (total of 3 BART and 3 blood sample collections per patient per visit).

Brachial artery reactivity studies will be conducted per following protocol:

* Equipment - Echocardiography system w/vascular software for 2-D imaging, Doppler and high-frequency vascular transducer.
* Initial image - Subject will be placed in a temperature-controlled room (22Cº). With subject positioned supine, left brachial artery will be imaged 5 cm above antecubital crease in longitudinal plane twice. Blood pressure and heart rate will be also measured.
* FMD - 12.5 cm blood pressure cuff will be placed above the antecubital fossa on left arm, baseline flow velocity will be obtained by pulsed Doppler. Thereafter, artery will be occluded by cuff inflation to 50 mm Hg above systolic pressure for 5 minutes and subsequently deflated. The longitudinal image will be obtained 1 min after cuff release.
* FMD w/NTG - 10 min after baseline study, FMD with NTG will be obtained. 0.4 mg sublingual NTG tablet will be given to subject and 4 min later, FMD imaging will be repeated as described above.
* Analysis - Photographic images of end-diastolic frames will be obtained. Images will be analyzed by 2 independent investigators blinded to the subject's identity and temporal sequence of images. Arterial diameter of the brachial artery in longitudinal plane from images where there is clear visualization of anterior and posterior intimal/lumen interface will be determined by caliper measurement. FMD quantified as a percent diameter change of the post-occlusion arterial diameter measurement relative to the mean of the 2 corresponding baseline measurements. Similar analysis will be performed for FMD following administration of NTG.

Lipid testing will be performed using the VAP® test and will include VLDL, LDL, HDL and IDL lipoprotein fractions as well as Triglycerides, Lipoprotein A, CRP and Homocysteine. Statistical analysis will be conducted as follows: group values for percent change in arterial diameter will be expressed as mean +/- SD. 2- tailed paired t-test will be used to compare changes in individual subjects. Two-tailed non-paired t-test will be used to compare values between groups. The analyses for FMD - lipid lowering correlation will be performed using a paired t test for parametrically distributed data and the Wilcoxon matched-pair signed rank test for nonparametrically distributed data to compare baseline data and changes in all variables at the end of the study within each group. The t test will used to compare the baseline characteristics between those receiving ezetimibe and those receiving placebo in all groups. Correlation between variables will be tested using both univariate and multitivariate analyses. The results will be presented as mean ± SD andmedian (25-75 percentiles).

ELIGIBILITY:
Inclusion Criteria:

* healthy adults over 18 yrs of age

Exclusion Criteria:

* presence of known metabolic syndrome
* as history of coronary artery disease
* hypertension
* diabetes
* cardiomyopathy
* tobacco use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ori Ben-Yehuda, MD, Principal Investigator — UCSD

RESULTS

PARTICIPANT FLOW:
Groups:
- Ezetimibe, Then Placebo: Participants first recieved ezetimibe, after a washout period of 2 weeks, they then received a placebo.
- Placebo, Then Ezetimibe: Participants first recieved a placebo, after a washout period of 2 weeks, they then received ezetimibe.
Period: First Intervention (2 Weeks)
Arm/Group | Ezetimibe, Then Placebo | Placebo, Then Ezetimibe
Started | 14 | 14
Completed | 10 | 12
Not Completed | 4 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Period: Washout (2 Weeks)
Arm/Group | Ezetimibe, Then Placebo | Placebo, Then Ezetimibe
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | Ezetimibe, Then Placebo | Placebo, Then Ezetimibe
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All subjects were randomized to ezetimibe or placebo, allowed a washout period, and then crossed over to the other arm. The demographic data is presented as all participants because the only data available at this time is the aggregated data and there is no access to the primary source data due to the age of this study.
Arm/Group | All Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Flow Mediated Dilation
Time Frame: before food, 3 hours postprandially and 6 hours postprandially
Measure: Median (Standard Deviation); unit: percent change
Groups:
- Placebo; Ezetimibe: Subjects were randomized to ezetimibe vs. placebo, allowed a washout period, and then crossed over to the other arm.
Arm/Group | Placebo | Ezetimibe
Number analyzed (Participants) | 22 | 22
percent change
  Before Food (0 hour) | 12.3 (4.5) | 11.6 (4.3)
  3 Hours Postprandially | 10.9 (5.5) | 11.1 (6.3)
  6 Hours Postprandially | 12.8 (4.3) | 13.9 (6.2)

2. Secondary Outcome: Lipid Profile- Change in LDL(Low Density Lipoprotein)
Time Frame: before food, 3 hours post prandial, 6 hours postprandial
Population: The results are reported for ezetimibe and placebo irrespective of order of administration, (there was a washout period of 4-6)
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Ezetimibe; Placebo: All Participants received both ezetimibe and placebo in cross over design.
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 22 | 22
mg/dl
  before food (0 hour) | 92 (24) | 102 (30)
  3 hour postprandial | 89 (22) | 104 (27)
  6 hour postprandial | 87 (23) | 101 (28)

ADVERSE EVENTS:
Time Frame: Through Study Completion (total of 8 weeks)
Arm/Group | Ezetimibe | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 2/28 | 0/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe (N=28) | Placebo (N=28)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes